CLINICAL TRIAL: NCT05466721
Title: HydrustomaC3 - Randomized Clinical Trial to Evaluate Safety and Efficacy of Innovative Medical Devices for Colostomy Patients
Brief Title: Evaluate Safety and Efficacy of Innovative Medical Devices for Colostomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hydrumedical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HydrustomaC3
Record Dates: First submitted 2022-06-29; First posted 2022-07-20 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Colostomy Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrustoma C3 (Experimental): The participant will use the Hydrustoma C3 devices for 14 days and then switch into the control device for another 14 days.
  Interventions: Device: Hydrustoma C3; Device: Coloplast Alterna
- Coloplast Alterna (Other): The participant will use the control devices for 14 days and then switch into the Hydrustoma C3 devices for another 14 days.
  Interventions: Device: Hydrustoma C3; Device: Coloplast Alterna

INTERVENTIONS:
Device: Hydrustoma C3 — The participant will use the device for 14 days.
Device: Coloplast Alterna — The participant will use the device for 14 days.

SUMMARY:
The surgical ostomy process happens when it is necessary to open an organ (such as the intestine) in order to maintain a communication channel with the external environment. The need for ostomy surgery can happen as a result of illness, genetic factors, or trauma. Despite the extensive improvements in colorectal surgery, in case there is a need for total or partial extraction and exteriorization of the large intestine (colostomy), it is often necessary to perform a stoma that connects the end of the preserved intestine to the skin, in which cases it is necessary to place a a colostomy bag for stool collection. Thus, there is a substantial number of patients who need to live with a permanent abdominal stoma that significantly affects their quality of life, implying significant changes, both physical and social. It will then be necessary for patients to adjust their daily routines in order to deal with stoma care.

The primary objective of this study is to evaluate the Hydrustoma C3 medical devices (plate C3, capsule C3, night bag C3) in terms of its efficacy and safety as colostomy devices. It is also a primary objective of this study to compare the health-related quality of life in patients with colostomy when using a control and Hydrustoma C3 devices.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* Male and Female patients;
* Adult aged ≥ 18;
* Descending and sigmoid colostomy created more than 3 months previously to the beginning of the study;
* Having formed stool and using a flat ostomy appliance;
* Able to understand the study procedures and fill questionaries;
* Able to apply and remove the ostomy device autonomously.

Exclusion Criteria:

* Repeated experiences of leakage with the usual ostomy device,
* Chronically liquid stools,
* Peristomal skin disorders,
* Known allergic reactions to components of the device,
* Receiving chemotherapy, radiation therapy or steroids in the previous month

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of the device (journal of capsule/bag changes) | 14 days
  Efficacy will be accessed by asking patients to record on a journal/diary, for each capsule/bag change, what was the reason for the change, and the occurrence and level of leakage.
Quality of life of the participant (Stoma Quality of Life questionnaire) | 14 days
  In order to compare stoma related quality of life in patients with colostomy when using a control device and the Hydrustoma C3 devices the Stoma Quality of Life questionnaire will be used. This questionnaire is composed of 20 questions. Example of question "I worry that the bag detaches.". All questions must be answered on a scale of 1 to 4, being 1 always and 4 never.
Adverse effects | 14 days
  Safety evaluations will be done by monitoring adverse events.
Safety of the device (Discolouration, Erosion, Tissue overgrowth score) | 14 days
  Safety evaluations will be done by monitoring the peristomal skin using the validated Ostomy Skin tool (DET score). The DET Score is calculated by examining the peristomal skin and evaluate the skin based on the descriptions in each of the 3 domains, discolouration (D), erosion (E) and tissue overgrowth (T); and assessing the size of the area affected in each of the 3 domains. The total score is (maximum 15) calculated by adding all of the subscores from each domain together.

SECONDARY OUTCOMES:
Satisfaction of the participant (questionnaire) | 14 days
  The patients will be asked to evaluate the medical device in terms of application, discretion of the device, stoma related noise, feelings of security (confidence) and overall satisfaction of use (including comfort and impact on body image). The questionnaire has 8 questions of multiple choice (example "Regarding the safety during usage of the devices, I feel: (1) very insecure; (2) moderately insecure; (3) Moderadately secure; (4) Very secure") and 1 open answer question.

CONTACTS AND LOCATIONS:
Overall Officials: Palmira Peixoto, Principal Investigator — Hospital de Braga; Paula Costa, Principal Investigator — Hospital Da Senhora Da Oliveira - Guimarães; Liliana Miranda, Principal Investigator — Hospital Centre Hospitalar de Trás-os-Montes e Alto Douro; Sara Costa, Principal Investigator — Centro Hospitalar de Entre o Douro e Vouga; Glória Gonçalves, Principal Investigator — Centro Hospitalar de Vila Nova de Gaia/Espinho; Carla Nunes, Principal Investigator — Centro Hospitalar do Tâmega e Sousa
Locations (6):
- Portugal (6):
  - Hospital Da Senhora Da Oliveira - Guimarães, Guimarães, Braga District
  - Hospital de Braga, Braga
  - Centro Hospitalar do Tâmega e Sousa, Penafiel
  - Centro Hospitalar de Entre o Douro e Vouga, Santa Maria da Feira
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, Vila Nova de Gaia
  - Centro Hospitalar de Trás-os-Montes e Alto Douro, Vila Real